CLINICAL TRIAL: NCT05925933
Title: Effect of High Protein Diet on Transcriptomic Regulations, Plasma Metabolomics, Hepatic and Pancreatic Fat Anatomy and Physiology in Asian Indians With Pre-diabetes
Brief Title: High Protein Diet on Transcriptomic, Metabolomics, Hepatic and Pancreatic Fat Anatomy and Physiology in Asian Indians With Pre-diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diabetes Foundation, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DFI/DST/2023
Record Dates: First submitted 2023-06-13; First posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Pre-diabetes
MeSH Terms: conditions — Glucose Intolerance | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Protein Diet (Experimental): High protein diet (carbohydrates 45%, protein 29%, and fat 26%) over 8-week periods. All assessments as done on day 1 will be repeated on day 60.
  Interventions: Other: Intervention
- Control Group (Other): Equicaloric normal diet (carbohydrates 60%, protein 15%, and fat 25%)
  Interventions: Other: Intervention

INTERVENTIONS:
Other: Intervention — high protein diet (carbohydrates 45%, protein 29%, and fat 26%) over 8-week periods.

SUMMARY:
Diabetes/ prediabetes is a substantial problem in India not only because it itself can be associated with morbidities such as coronary artery disease but also because it is a point of importance for the prevention of other diseases. It is not clear if a high protein calorie diet in the Indian population associated with a heightened tendency for prediabetes, metabolic syndrome, atherosclerosis and dysmetabolic state etc. could, besides lifestyle factors, be related to diet, or interaction between the two. The analysis of whole blood transcriptomes and plasma metabolomics profiles may be a potentially useful tool for the assessment of metabolic health status. The proposed study is the first to perform a detailed gene expression profiling with the use of next-generation sequencing technology to assess the differences in molecular mechanisms in the peripheral blood of subjects with prediabetes.

DETAILED DESCRIPTION:
This study will be conducted at the outpatient department of the National Diabetes, Obesity and Cholesterol Foundation (N-DOC), Diabetes Foundation (India) (DFI)and Fortis-C-DOC, Centre of Excellence for Diabetes, Metabolic Diseases and Endocrinology, New Delhi, India.

Experimental Protocol: In this study, a total of 60 subjects with pre-diabetes and 60 age and body mass index, and gender-matched controls (age 18-40 years) will be recruited. They will be randomized to an equicaloric normal diet (carbohydrates 60%, protein 15%, and fat 25%) or a high protein diet (carbohydrates 45%, protein 29%, and fat 26%) over 8-week periods. All assessments as done on day 1 will be repeated at day 60.

ELIGIBILITY:
Exclusion Criteria:

* Acute infections and advanced end-organ damage.
* History of hepatitis or pancreatitis, abnormal liver and renal function tests.
* Recent (<3 months) changes in weight (≥5%) and/or weight changing medications.
* Subjects with metallic implants, pacemaker leads, radioactive seeds or surgical staples in the body.

Inclusion Criteria

Cases:

* Age 18 to 50 years. Subjects with pre-diabetes on oral glucose tolerance test (OGTT)
* Fasting blood glucose≥100mg/dl and <126 mg/dl or 2-h plasma glucose ≥140mg/dl and <200mg/dl (after ingestion of 75 grams of anhydrous oral glucose) or both.

Controls:

* Age 18 to 50 years. Normoglycemia by OGTT
* Fasting blood glucose <100mg/dl and 2-h plasma glucose <140mg/dl (after ingestion of 75 gram of anhydrous oral glucose).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index | 6 Months
  BMI will be calculated by using formula weight (Kg)/height (m2).
Body Fat | 2 MONTHS
  Body estimations will be done by DEXA Scan
Liver Fat | 2 Months
  Liver fat will be done by MRI Scan
Next Generation sequencing | 06 MONTHS
Pancreatic fat | 06 MONTHS
  Pancreatic fat estimation will be done by MRI
RNA Extraction | 06 MONTHS
Metabolomics profile | 06 MONTHS

IPD SHARING:
Plan to Share IPD: No
In this study a total of 60 subjects with pre-diabetes and 60 age and body mass index, and gender matched controls (age 18-40 years) will be recruited. They will be randomized to an equicaloric normal diet or high protein diet over 8-week periods. All assessments as done on day 1 will be repeated on day 60.